CLINICAL TRIAL: NCT07317050
Title: Aprotinin Treatment of Acute Respiratory Distress Syndrome: a Multicenter, Double-blind, Placebo-controlled, Phase III Trial
Brief Title: Clinical Trial With Aprotinin in the Acute Respiratory Distress Syndrome Treatment
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion del Hospital Nacional de Paraplejicos para la Investigacion y la Integracion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICI24/00011; 2025-520826-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: Acute Respiratory Distress Syndrome (ARDS); Inhaled Aprotinin; Phase III Clinical Trial; Ventilator-free days; Pulmonary Function; Inflammatory Biomarkers
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Aprotinin; Inhalation; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Phase III, multicentre, double-blind, randomized, parallel-group clinical trial evaluating the efficacy and safety of inhaled aprotinin versus placebo in adult patients with moderate or severe ARDS.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled Aprotinin Group (Experimental): Patients in this Experimental Group will receive inhaled aprotinin as an adjunctive therapy to standard supportive care for ARDS. Treatment is administered four times daily for 6 consecutive days. All patients continue to receive standard supportive care according to local practice.
  Interventions: Drug: Aprotinin (inhaled)
- Inhaled Placebo Group (Placebo Comparator): Patients in this Control Group will receive inhaled placebo (sodium chloride) as an adjunctive therapy to standard supportive care for ARDS. Administration schedule matches the experimental group, four times daily for 6 consecutive days. All patients continue to receive standard supportive care according to local practice.
  Interventions: Drug: Placebo (Sodium Chloride)

INTERVENTIONS:
Drug: Aprotinin (inhaled) — Inhaled aprotinin, diluted in 0.9% sodium chloride, is administrated via nebulization through an endotracheal or tracheostomy tube. The dose is 500 UI every 6 hours (totaling 2,000 UI/day) for six consecutive days. Each administration consists of a nebulized inhalation lasting no less than six minutes, with four inhalations delivered per day. Nebulization is performed using Aerogen® Solo vibrating mesh nebulizers to maintain a closed ventilatory circuit. The device produces aerosol particles with a median diameter of 2-10 µm; 30-50% of these aggregates reach diameters of 50-100 µm. Administration follows pharmacy blinding procedures. All patients receive standard supportive care according to local practice.
  Arms: Inhaled Aprotinin Group
Drug: Placebo (Sodium Chloride) — Placebo (sodium chloride) is administered by inhalation via endotracheal or tracheostomy tube using the Aerogen® Solo vibrating mesh nebulizer, four times daily for six consecutive days. It is delivered following the same dosing schedule, device specifications, and administration procedures as the active treatment. Administration follows pharmacy blinding procedures to maintain double-blind conditions. All patients receive standard supportive care according to local practice.
  Arms: Inhaled Placebo Group

SUMMARY:
This is a multicentre, double-blind, placebo-controlled Phase III randomized clinical trial designed to evaluate the efficacy and safety of inhaled aprotinin in adult patients with moderate or severe acute respiratory distress syndrome (ARDS). A total of 156 critically ill patients admitted to intensive care units will be randomized to receive either inhaled aprotinin or placebo in addition to standard supportive care. The primary objective is to determine whether aprotinin improves clinical outcomes based on a composite endpoint of mortality and ventilator-free days at 28 days.

DETAILED DESCRIPTION:
This study is a nation-wide, multicentre, double-blind, placebo-controlled, Phase III randomized clinical trial designed to investigate the efficacy and safety of inhaled aprotinin in adult patients diagnosed with moderate or severe acute respiratory distress syndrome (ARDS). ARDS is a heterogeneous acute inflammatory lung syndrome characterized by diffuse alveolar damage, increased vascular permeability, alveolar and interstitial edema, and severe hypoxemic respiratory failure. Despite advances in supportive care, no specific pharmacological therapy has demonstrated proven benefit.

Aprotinin is a broad-spectrum serine protease inhibitor that targets the kallikrein-kinin system and attenuates systemic inflammatory responses, including reductions in pro-inflammatory cytokines and matrix metalloproteinases (MMPs). Experimental and clinical data suggest that MMP overexpression contributes to tissue damage, coagulation abnormalities, and impaired lung repair, representing a potential therapeutic target in ARDS. Inhaled aprotinin has been used clinically in patients with respiratory conditions, including COVID-19 and chronic pulmonary disease, with no reported adverse events via this route of administration.

In this trial, 156 ICU patients with moderate or severe ARDS will be enrolled and randomized in a 1:1 ratio to receive either inhaled aprotinin or placebo, both administered alongside standard supportive care. The aprotinina dosing regimen will be four inhaled doses of 500 KIU every six hours (total 2,000 KIU/day), selected to achieve effective local pulmonary concentrations while minimizing systemic exposure. The primary endpoint is a composite of mortality and ventilator-free days at 28 days among survivors. Secondary outcomes include ICU and hospital mortality, duration of mechanical ventilation, and other clinically relevant respiratory and functional endpoints. Detailed study procedures, dosing, and administration are described in the study protocol.

All study procedures will be conducted under a double-blind design. Patients will be prospectively followed for clinical outcomes during their ICU and hospital stay according to prespecified assessment timepoints. A Data Monitoring Committee (DMC) composed of independent clinical experts will periodically review safety and efficacy data, ensuring the protection of participants and the scientific validity of the study. The estimated study duration is four years, from September 2025 to September 2029.

ELIGIBILITY:
Inclusion Criteria:

Each potential participant must satisfy all of the following criteria to be enrolled in the study:

1. Diagnosed with moderate or severe Acute Respiratory Distress Syndrome (ARDS) according to the Berlin definition (ARDS Definition Task Force 2012):

   * Acute onset of respiratory failure within 1 week of a known clinical insult or new/worsening respiratory symptoms.
   * Respiratory failure not fully explained by cardiac failure or fluid overload; objective evaluation of cardiac failure or fluid overload is required if ARDS risk factors are absent.
   * Radiographic abnormalities on chest X-ray or CT scan: bilateral opacities not fully explained by effusions, nodules, masses, or lobar/segmental collapse.
   * Hypoxemia:

     * Moderate ARDS: PaO₂/FiO₂ >100 mmHg and ≤200 mmHg with Positive End-Expiratory Pressure (PEEP) ≥5 cmH₂O.
     * Severe ARDS: PaO₂/FiO₂ ≤100 mmHg with PEEP ≥5 cmH₂O.
2. Radiographic and hypoxemia criteria must occur within the same 24-hour period. ARDS onset is defined as the time when the last of these two criteria is met.
3. First dose of study drug planned within 48 hours of moderate or severe ARDS diagnosis.
4. Intubated and receiving mechanical ventilation.
5. Age ≥18 years.
6. Women of childbearing potential must have a negative serum pregnancy test during screening and a negative urine pregnancy test at study start. Female subjects of childbearing potential and male subjects with partners of childbearing potential must agree to use an effective contraceptive method from consent until 30 days after study drug administration.

Exclusion Criteria:

Any potential participant who meets any of the following criteria will be excluded from participating in the study:

1. Pregnant or lactating women, or positive/indeterminate pregnancy test (serum or urine).
2. Simultaneous participation in another pharmacotherapy protocol.
3. Life expectancy <24 hours.
4. Clinical condition in which, in the investigator's opinion, ventilator withdrawal is extremely unlikely (e.g., motor neuron disease, Duchenne muscular dystrophy, rapidly progressive interstitial lung disease).
5. Severe chronic obstructive pulmonary disease requiring long-term home oxygen or mechanical ventilation (noninvasive or tracheostomy), except Continuous Positive Airway Pressure (CPAP) or Bilevel Positive Airway Pressure (BiPAP) used solely for sleep-related respiratory disorders.
6. Congestive heart failure defined as New York Heart Association (NYHA) class IV.
7. Acute left ventricular failure.
8. Severe hepatic impairment (Child-Pugh class C).
9. Prior interferon therapy.
10. Known hypersensitivity to natural or recombinant IFN beta or any excipients.
11. Receiving renal dialysisfor chronic renal failure.
12. Receiving extracorporeal membrane oxygenation (ECMO), high-frequency oscillatory ventilation, or any form of extracorporeal pulmonary support.
13. Mechanical ventilation, (invasive or noninvasive, excluding CPAP alone), for more than 48 hours before ARDS diagnosis. Noninvasive ventilation must be applied continuously for at least 12 hours/day during those 48 hours.
14. Burns covering ≥15% total body surface.
15. Women with positive pregnancy test at screening (serum) or study start (urine); lactating subjects; subjects planning pregnancy within 1 month after the study (including male partners).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Ventilator-Free Days (VFD) in patients with moderate or severe ARDS | From first dose up to Day 28
  Number of days a patient is free from invasive mechanical ventilation (DLVI) within 28 days after first dose. A patient is considered ventilator-free after two consecutive calendar days of unassisted breathing. This outcome will be used to assess the efficacy of inhaled aprotinin compared with placebo.

SECONDARY OUTCOMES:
Number of participants with at least one treatment-emergent adverse event | From first dose up to Day 180
  Incidence, severity, and relationship to treatment of adverse events (AEs), coded according to MedDRA (Medical Dictionary for Regulatory Activities), in treated participants. This outcome evaluates the safety profile of aprotinin compared with placebo.
Proportion of patients who die from any cause within 28, 90, or 180 days after receiving first dose of study treatment. | At Day 28, Day 90, and Day 180
  All-Cause Mortality.
Number of days free from ICU or hospital | From first dose up to Day 28
  Total number of days a patient remains outside the intensive care unit (ICU) and outside the hospital within 28 days after receiving first dose of study treatment.
Number of days on renal or vasoactive support within 28 days after first dose | From first dose up to Day 28
  Total number of days a patient requires renal replacement therapy or vasoactive support within 28 days after receiving first dose of study treatment.
Sequential Organ Failure Assessment (SOFA) score | From Day 1 up to Day 28
  Sequential Organ Failure Assessment (SOFA) score evaluated daily from Day 1 to Day 14, and on Days 21 and 28.
PaO₂/FiO₂ ratio during mechanical ventilation | From Day 1 up to Day 28
  Daily evaluation of the arterial oxygen partial pressure to inspired oxygen fraction (PaO₂/FiO₂) ratio during mechanical ventilation as an indicator of pulmonary function improvement in patients receiving study treatment.
Plasma inflammatory biomarkers | Day 1 and Day 5
  Measurement of plasma levels of selected pro- and anti-inflammatory cytokines (GM-CSF, IFN-α, IFN-γ, IL-1α, IL-1β, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, IL-17A, TNF-α), chemokines (IP-10/CXCL10, MCP-1/CCL2, MIP-1α/CCL3, MIP-1β/CCL4), and cell adhesion/response markers (ICAM-1, CD62E/E-selectin, CD62P/P-selectin) in plasma on Day 1 and Day 5 in all participants receiving study treatment. Evaluates the effect of aprotinina on systemic inflammation.
Pulmonary biomarkers in bronchial and plasma samples | Day 1 and Day 5
  Determination of granular proteins, bradykinin, and kallikreins in bronchial brush and plasma samples on Day 1 and Day 5 as exploratory markers of pulmonary response and treatment effect of aprotinin.
Plasma aprotinin levels | Day 1 and Day 5
  Measurement of plasma aprotinin concentrations on Day 1 and Day 5 in all participants receiving study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario de Ciudad Real, Ciudad Real, Ciudad Real, Spain

IPD SHARING:
Plan to Share IPD: No